CLINICAL TRIAL: NCT05042622
Title: Innovative Solutions to Organ-substituting Technologies in the Treatment of Heart and Pulmonary Failure
Brief Title: Organ-substituting Technologies in the Treatment of Heart and Pulmonary Failure
Acronym: OST
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Research Center for Cardiac Surgery, Kazakhstan (Other)
Collaborators: Ministry of Education and Science, Republic of Kazakhstan (Other Government)
Responsible Party: Principal Investigator, Timur Lesbekov, Head of the Department of Cardiac Surgery, National Research Center for Cardiac Surgery, Kazakhstan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: version 1.1
Record Dates: First submitted 2021-08-20; First posted 2021-09-13 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Acute Respiratory Distress Syndrome; Septic Shock; Sepsis
Keywords: Organ-substituting technologies; Heart failure; Pulmonary failure; Sepsis; Extracorporeal membrane oxygenation; Adsorber
MeSH Terms: conditions — Respiratory Distress Syndrome; Shock, Septic; Sepsis; Heart Failure

STUDY DESIGN:
Intervention Model Description: Study Design Study Type: Interventional (Clinical Trial) Estimated Enrollment: 90 Participants Allocation: randomized Interventional Model: Parallel assignment Masking: None (Open Label)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cytokine adsorber patients on ECMO (Experimental): Cytokine adsorber filter will be installed into the (hemodialysis or cardiopulmonary bypass (CPB) (15 patients on ECMO)
  Interventions: Device: Cytokine adsorber filter
- Cytokine adsorber patients with sepsis (Experimental): Cytokine adsorber filter will be installed into the (hemodialysis or cardiopulmonary bypass (CPB) (15 patients with sepsis)
  Interventions: Device: Cytokine adsorber filter
- Extracorporeal hemoperfusion cartridge patients on ECMO (Experimental): Extracorporeal hemoperfusion cartridge will be installed into the (hemodialysis or cardiopulmonary bypass (CPB) (15 patients on ECMO)
  Interventions: Device: Extracorporeal hemoperfusion cartridge
- Extracorporeal hemoperfusion cartridge patients with sepsis (Experimental): Extracorporeal hemoperfusion cartridge will be installed into the (hemodialysis or cardiopulmonary bypass (CPB) (15 patients with sepsis)
  Interventions: Device: Extracorporeal hemoperfusion cartridge
- Control (subgroups)1 (No Intervention): No filter will be installed into the ECMO in this study group (15 patients)
- Control (subgroups) 2 (No Intervention): No filter will be installed into the patient with sepsis (15 patients)

INTERVENTIONS:
Device: Cytokine adsorber filter — • Intervention group #1 a cytokine adsorber will be used (30 patients): patients on ECMO - subgroup A; septic patients - subgroup B.
  Arms: Cytokine adsorber patients on ECMO; Cytokine adsorber patients with sepsis
Device: Extracorporeal hemoperfusion cartridge — • Intervention group #2 an extracorporeal hemoperfusion cartridge will be used (30 patients): patients on ECMO - subgroup C, septic patients - subgroup D.
  Arms: Extracorporeal hemoperfusion cartridge patients on ECMO; Extracorporeal hemoperfusion cartridge patients with sepsis

SUMMARY:
The implementation of this project will improve the effectiveness of surgical treatment and reduce the level of complications and mortality among patients with heart failure and heart failure in the terminal stage.

The goal of the study. Improvement of organ-substituting technologies in the treatment of heart and respiratory failure.

Objectives of the study. Objective 1. To study the restoration of organ function during implantation of extracorporeal membrane oxygenation (ECMO), as an organ replacement, in cardiac and / or respiratory failure.

Objective 2. To study the results of applying organ-substituting technologies in the treatment of sepsis.

DETAILED DESCRIPTION:
The implementation of this project will improve the effectiveness of surgical treatment and reduce the level of complications and mortality among patients with heart failure and heart failure in the terminal stage.

2.2. The goal of the program. Improvement of organ-substituting technologies in the treatment of heart and respiratory failure.

2.3. Objectives of the program. Objective 1. To study the restoration of organ function during implantation of extracorporeal membrane oxygenation (ECMO), as an organ replacement, in cardiac and/or respiratory failure.

Subtask 1.1. Evaluation of the recovery of organ function during ECMO using extracorporal hemo correction procedure.

Subtask 1.2. Evaluation of the normalization of the organism's immune response and restoration of organ function when conducting ECMO using the extracorporeal cytokine adsorber.

Subtask 1.3. Evaluation of the normalization of the organism's immune response and restoration of organ function when conducting ECMO using the extracorporeal hemoperfusion cartridge.

Objective 2. To study the results of applying organ-substituting technologies in the treatment of sepsis.

Subtask 2.1. Assessment of the recovery of organ function in the application of extracorporal hemo correction in septic patients.

Subtask 2.2. Evaluation of the normalization of the organism immune response and restoration of organ function when using the extracorporeal cytokine adsorber in septic patients.

Subtask 2.3. Evaluation of the normalization of the organism's immune response and restoration of organ function when using the extracorporeal hemoperfusion cartridge.

In this study, will be developed methods to restore the function of affected organs after implantation of ECMO and patients with sepsis in combination with extracorporeal hem correction, which will improve the results of surgical treatment of patients with end-cardiac and respiratory failure.

New methods developed to restore the function of affected organs after implantation of mechanical support devices and patients with sepsis will be of great importance both for Kazakhstan and for countries with similar categories of patients, which will improve the efficiency of surgical treatment and reduce the level of complications and mortality.

Clinical research data will form the basis of practical protocols for extracorporeal membrane oxygenation (ECMO) and patients with sepsis, which will improve organ repair, reduce postoperative complications, improve quality of life and reduce mortality after surgery.

Research methods and ethical issues Patients before implantation of ECMO and/or patients with sepsis will be enrolled in the study after giving a written, signed informed consent.

The participants will be randomized into 3 groups:

* Intervention group #1 a cytokine adsorber will be used (30 patients): patients on ECMO - subgroup A; septic patients - subgroup B.
* Intervention group #2 an extracorporeal hemoperfusion cartridge will be used (30 patients): patients on ECMO - subgroup C, septic patients - subgroup D.
* Control group #3 without using extracorporeal adsorber (30 patients): patients on ECMO subgroup - E, septic patients - subgroup F.

The investigators will collect demographic, clinical, and laboratory data about patients before, during, and after the operation The incidence of early cellular or humoral rejection, length of ventilation, ICU and hospital stay, the use of vasopressors and inotropes in the perioperative period, and incidence of perioperative complications and survival will be documented.

The level of cytokines (IL-1, IL-6, IL-8, IL-10, tumor necrosis factor-alfa) and complements before, during, and after the use of ECMO, patients with sepsis will be determined if the investigators find the relevant differences between the two groups in clinical variables.

Study Design Study Type: Interventional (Clinical Trial) Estimated Enrollment: 90 Participants Allocation: randomized Interventional Model: Parallel assignment Masking: None (Open Label)

ELIGIBILITY:
Inclusion Criteria:

-

ICU patients with ECMO:

* Hemodynamic support with vasopressors
* Procalcitonin level ≥ 1 ng/ml
* Invasive hemodynamic monitoring
* Written informed content

ICU patients with the septic shock of medical origin:

* Signs of hypoperfusion: serum lactate >2 mmol/L, low central venous oxygen saturation (ScvO2) (<70%) or high ScvO2 (>85%), metabolic acidosis, oligo-anuria, high venous-to-arterial CO2-gap (dCO2 >6 mm Hg)
* Hemodynamic support with vasopressors
* Procalcitonin level ≥ 1 ng/ml
* Invasive hemodynamic monitoring
* Written informed content

Exclusion Criteria:

* ICU patients with ECMO:

  * age < 18 years
  * acute liver or kidney failure straight before transplantation
  * the patient declines to participate in the study

ICU patients with the septic shock of medical origin:

* Patients under 18 years
* Pregnancy (bHCG test positivity)
* Surgical intervention in context with the septic insult New York Heart Association IV heart failure
* Acute coronary syndrome
* Acute hematological malignancies
* Immunosuppression, systemic steroid therapy (>10mg prednisolone/day)
* Human immunodeficiency virus infection (HIV) and active AIDS
* Patients with donated organs
* Thrombocytopenia (<20.000/ml)
* More than 10%-of body surface area with third-degree burn

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Difference of Cytokine response - ECMO patients | 6-24 hours
  Level of pro- and anti-inflammatory cytokines (IL-1, IL-6, IL-8, IL-10, tumor necrosis factor-alfa) before initiation of ECMO, 2 hours after initiation ECMO support, at explantation of ECMO support, 6-12-24 hours after explantation of ECMO support.
Difference of Cytokine response - Patients with septic shock | 24-48 hours of septic shock
  Level of procalcitonin, Level of C-reactive protein, Level of interleukin-1, Level of interleukin-6, Level of interleukin-8, Level of interleukin-10, Level of Tumor Necrosis Factor- αinterleukin-8, interleukin-10, Tumor Necrosis Factor- α at 24, 48 hours.

SECONDARY OUTCOMES:
Inflammatory reaction - Patients with septic shock | 6-24 hours
  Level of C reactive protein (CRP), white blood cells and procalcitonin immediately after induction of anesthesia, before initiation of adsorber, 2 hours after initiation of adsorber, at termination of adsorber, 6-12-24 hours after wean of adsorber.
Ventilator free days (VFD) - ECMO patients | 30 days
  ventilator days. VFD=0, if the patient dies in the first 30 days after randomization
Time to extubation from ventilation and explantation from ECMO - ECMO patients | 30 days
  Time to extubation from ventilation and explantation from ECMO. Death under ventilation and/or ECMO will be analyzed as a competing event. The time will be censored at the time of last visit for surviving patients under ventilation and/or ECMO.
Difference of d-dimers - ECMO patients | 24, 48, 72 hours
  Comparison to enrollment or between 3 groups at 24, 48, 72 h
Difference of Serum lactate - ECMO patients | 24, 48, 72 hours
  Comparison to enrollment or between 3 groups at 24, 48, 72 h
SOFA-Score - ECMO patients | 24, 48, 72 hours
  Sequential Organ Failure Assessment Score at 24, 48, 72 h (values from 6 to 24, where the higher values explain higher disease severity)
serious adverse device effects - ECMO patients | 30 days
  serious complications or malfunctions related to the CytoSorb device
adverse event of special interest: air in the ECMO system - ECMO patients | 30 days
  unintended air in the ECMO system during operation of the device
adverse event of special interest: blood-clotting in the ECMO system | 30 days
  unintended blood-clotting in the ECMO system during operation of the device
adverse event of special interest: bleeding complications - ECMO patients | 30 days
  major bleeding events
Difference of serum interleukin-6 level - Patients with septic shock | 48, 72 hours
  Comparison to enrollment or between 3 groups at 48, 72 h
Difference of serum interleukin-1β level - Patients with septic shock | 24, 48, 72 hours
  Comparison to enrollment or between 3 groups at 24, 48, 72 h
Difference of serum interleukin-10 level - Patients with septic shock | 24, 48, 72 hours
  Comparison to enrollment or between 3 groups at 24, 48, 72 h
Difference of serum procalcitonin level - Patients with septic shock | 24, 48, 72 hours
  Comparison to enrollment or between 3 groups at 24, 48, 72 h

OTHER OUTCOMES:
Overall survival time | 30 days
  Overall survival time, defined as time from randomization to death. The time will be censored at the time of last visit for surviving patients.
Days on intensive care unit (ICU) | 30 days
  Days on intensive care unit (ICU)
Vasopressor dosage | 24, 48, 72 hours
  Vasopressor dosage of adrenaline, noradrenaline, vasopressin, and dobutamine at 24, 48,72 h
Fluid substitution and fluid balance | 24, 48, 72 hours
  Total fluid[ml] substitution and fluid balance [ml] at 24, 48, 72 h
Length of hospital stay | up to 1 months
  Days at hospital
Mortality | First 72 hours
  The period of occurrence of mortality

CONTACTS AND LOCATIONS:
Overall Officials: Timur Lesbekov, PhD, MD, Principal Investigator — National research Center for Cardiac Surgery JSC
Locations (1):
- National Research Center for Cardiac Surgery, Astana, Kazakhstan

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 01.01.2021 - 31.12.2023
Access Criteria: All patients will receive voluntary informed consent of the established sample with permission to use clinical data for scientific purposes. In addition, the study will be strictly controlled by researchers for the absence of plagiarism, falsification and fabrication of data in order to achieve the most ethical conduct of the study. The obtained patient data will be kept strictly confidential, ensuring privacy by strictly limited access to data, de-identification of data and destruction after the end of the study.
URL: http://heartcenter.kz

REFERENCES:
- [Background] Venet F, Lukaszewicz AC, Payen D, Hotchkiss R, Monneret G. Monitoring the immune response in sepsis: a rational approach to administration of immunoadjuvant therapies. Curr Opin Immunol. 2013 Aug;25(4):477-83. doi: 10.1016/j.coi.2013.05.006. Epub 2013 May 28. PMID 23725873
- [Result] Hunt SA. Taking heart--cardiac transplantation past, present, and future. N Engl J Med. 2006 Jul 20;355(3):231-5. doi: 10.1056/NEJMp068048. No abstract available. PMID 16855261
- [Result] Hunt SA, Haddad F. The changing face of heart transplantation. J Am Coll Cardiol. 2008 Aug 19;52(8):587-98. doi: 10.1016/j.jacc.2008.05.020. PMID 18702960
- [Result] Lund LH, Edwards LB, Kucheryavaya AY, Benden C, Christie JD, Dipchand AI, Dobbels F, Goldfarb SB, Levvey BJ, Meiser B, Yusen RD, Stehlik J; International Society of Heart and Lung Transplantation. The registry of the International Society for Heart and Lung Transplantation: thirty-first official adult heart transplant report--2014; focus theme: retransplantation. J Heart Lung Transplant. 2014 Oct;33(10):996-1008. doi: 10.1016/j.healun.2014.08.003. Epub 2014 Aug 14. No abstract available. PMID 25242124
- [Result] Banner NR, Thomas HL, Curnow E, Hussey JC, Rogers CA, Bonser RS; Steering Group of the United Kingdom Cardiothoracic Transplant Audit. The importance of cold and warm cardiac ischemia for survival after heart transplantation. Transplantation. 2008 Aug 27;86(4):542-7. doi: 10.1097/TP.0b013e31818149b9. PMID 18724223
- [Result] Russo MJ, Iribarne A, Hong KN, Ramlawi B, Chen JM, Takayama H, Mancini DM, Naka Y. Factors associated with primary graft failure after heart transplantation. Transplantation. 2010 Aug 27;90(4):444-50. doi: 10.1097/TP.0b013e3181e6f1eb. PMID 20622755
- [Result] Rihal CS, Naidu SS, Givertz MM, Szeto WY, Burke JA, Kapur NK, Kern M, Garratt KN, Goldstein JA, Dimas V, Tu T; Society for Cardiovascular Angiography and Interventions (SCAI); Heart Failure Society of America (HFSA); Society for Thoracic Surgeons (STS); American Heart Association (AHA); American College of Cardiology (ACC). 2015 SCAI/ACC/HFSA/STS Clinical Expert Consensus Statement on the Use of Percutaneous Mechanical Circulatory Support Devices in Cardiovascular Care (Endorsed by the American Heart Association, the Cardiological Society of India, and Sociedad Latino Americana de Cardiologia Intervencion; Affirmation of Value by the Canadian Association of Interventional Cardiology-Association Canadienne de Cardiologie d'intervention). J Card Fail. 2015 Jun;21(6):499-518. doi: 10.1016/j.cardfail.2015.03.002. PMID 26036425
- [Result] Mugford M, Elbourne D, Field D. Extracorporeal membrane oxygenation for severe respiratory failure in newborn infants. Cochrane Database Syst Rev. 2008 Jul 16;(3):CD001340. doi: 10.1002/14651858.CD001340.pub2. PMID 18646070
- [Result] Stretch R, Sauer CM, Yuh DD, Bonde P. National trends in the utilization of short-term mechanical circulatory support: incidence, outcomes, and cost analysis. J Am Coll Cardiol. 2014 Oct 7;64(14):1407-15. doi: 10.1016/j.jacc.2014.07.958. PMID 25277608
- [Result] McCarthy FH, McDermott KM, Kini V, Gutsche JT, Wald JW, Xie D, Szeto WY, Bermudez CA, Atluri P, Acker MA, Desai ND. Trends in U.S. Extracorporeal Membrane Oxygenation Use and Outcomes: 2002-2012. Semin Thorac Cardiovasc Surg. 2015 Summer;27(2):81-8. doi: 10.1053/j.semtcvs.2015.07.005. Epub 2015 Jul 22. PMID 26686427
- [Result] Maxwell BG, Powers AJ, Sheikh AY, Lee PH, Lobato RL, Wong JK. Resource use trends in extracorporeal membrane oxygenation in adults: an analysis of the Nationwide Inpatient Sample 1998-2009. J Thorac Cardiovasc Surg. 2014 Aug;148(2):416-21.e1. doi: 10.1016/j.jtcvs.2013.09.033. Epub 2013 Nov 1. PMID 24183903
- [Result] Tramm R, Ilic D, Davies AR, Pellegrino VA, Romero L, Hodgson C. Extracorporeal membrane oxygenation for critically ill adults. Cochrane Database Syst Rev. 2015 Jan 22;1(1):CD010381. doi: 10.1002/14651858.CD010381.pub2. PMID 25608845
- [Result] Chang CH, Chen HC, Caffrey JL, Hsu J, Lin JW, Lai MS, Chen YS. Survival Analysis After Extracorporeal Membrane Oxygenation in Critically Ill Adults: A Nationwide Cohort Study. Circulation. 2016 Jun 14;133(24):2423-33. doi: 10.1161/CIRCULATIONAHA.115.019143. Epub 2016 May 19. PMID 27199466
- [Result] Feldman D, Pamboukian SV, Teuteberg JJ, Birks E, Lietz K, Moore SA, Morgan JA, Arabia F, Bauman ME, Buchholz HW, Deng M, Dickstein ML, El-Banayosy A, Elliot T, Goldstein DJ, Grady KL, Jones K, Hryniewicz K, John R, Kaan A, Kusne S, Loebe M, Massicotte MP, Moazami N, Mohacsi P, Mooney M, Nelson T, Pagani F, Perry W, Potapov EV, Eduardo Rame J, Russell SD, Sorensen EN, Sun B, Strueber M, Mangi AA, Petty MG, Rogers J; International Society for Heart and Lung Transplantation. The 2013 International Society for Heart and Lung Transplantation Guidelines for mechanical circulatory support: executive summary. J Heart Lung Transplant. 2013 Feb;32(2):157-87. doi: 10.1016/j.healun.2012.09.013. No abstract available. PMID 23352391
- [Result] Khwannimit B, Bhurayanontachai R. The direct costs of intensive care management and risk factors for financial burden of patients with severe sepsis and septic shock. J Crit Care. 2015 Oct;30(5):929-34. doi: 10.1016/j.jcrc.2015.05.011. Epub 2015 May 20. PMID 26051981
- [Result] Iskander KN, Osuchowski MF, Stearns-Kurosawa DJ, Kurosawa S, Stepien D, Valentine C, Remick DG. Sepsis: multiple abnormalities, heterogeneous responses, and evolving understanding. Physiol Rev. 2013 Jul;93(3):1247-88. doi: 10.1152/physrev.00037.2012. PMID 23899564
- [Result] Kwan A, Hubank M, Rashid A, Klein N, Peters MJ. Transcriptional instability during evolving sepsis may limit biomarker based risk stratification. PLoS One. 2013;8(3):e60501. doi: 10.1371/journal.pone.0060501. Epub 2013 Mar 27. PMID 23544148
- [Result] Akira S, Uematsu S, Takeuchi O. Pathogen recognition and innate immunity. Cell. 2006 Feb 24;124(4):783-801. doi: 10.1016/j.cell.2006.02.015. PMID 16497588
- [Result] Hotchkiss RS, Monneret G, Payen D. Sepsis-induced immunosuppression: from cellular dysfunctions to immunotherapy. Nat Rev Immunol. 2013 Dec;13(12):862-74. doi: 10.1038/nri3552. Epub 2013 Nov 15. PMID 24232462
- [Result] Laszlo I, Trasy D, Molnar Z, Fazakas J. Sepsis: From Pathophysiology to Individualized Patient Care. J Immunol Res. 2015;2015:510436. doi: 10.1155/2015/510436. Epub 2015 Jul 15. PMID 26258150
- [Result] Cruz DN, Antonelli M, Fumagalli R, Foltran F, Brienza N, Donati A, Malcangi V, Petrini F, Volta G, Bobbio Pallavicini FM, Rottoli F, Giunta F, Ronco C. Early use of polymyxin B hemoperfusion in abdominal septic shock: the EUPHAS randomized controlled trial. JAMA. 2009 Jun 17;301(23):2445-52. doi: 10.1001/jama.2009.856. PMID 19531784
- [Result] Bellomo R, Baldwin I, Ronco C. Extracorporeal blood purification therapy for sepsis and systemic inflammation: its biological rationale. Contrib Nephrol. 2001;(132):367-74. doi: 10.1159/000060105. PMID 11395904
- [Result] Namas RA, Namas R, Lagoa C, Barclay D, Mi Q, Zamora R, Peng Z, Wen X, Fedorchak MV, Valenti IE, Federspiel WJ, Kellum JA, Vodovotz Y. Hemoadsorption reprograms inflammation in experimental gram-negative septic peritonitis: insights from in vivo and in silico studies. Mol Med. 2012 Dec 20;18(1):1366-74. doi: 10.2119/molmed.2012.00106. PMID 22751621
- [Result] Peng ZY, Carter MJ, Kellum JA. Effects of hemoadsorption on cytokine removal and short-term survival in septic rats. Crit Care Med. 2008 May;36(5):1573-7. doi: 10.1097/CCM.0b013e318170b9a7. PMID 18434884
- [Result] Peng ZY, Wang HZ, Carter MJ, Dileo MV, Bishop JV, Zhou FH, Wen XY, Rimmele T, Singbartl K, Federspiel WJ, Clermont G, Kellum JA. Acute removal of common sepsis mediators does not explain the effects of extracorporeal blood purification in experimental sepsis. Kidney Int. 2012 Feb;81(4):363-9. doi: 10.1038/ki.2011.320. Epub 2011 Sep 14. PMID 21918497
- [Result] Kellum JA, Venkataraman R, Powner D, Elder M, Hergenroeder G, Carter M. Feasibility study of cytokine removal by hemoadsorption in brain-dead humans. Crit Care Med. 2008 Jan;36(1):268-72. doi: 10.1097/01.CCM.0000291646.34815.BB. PMID 18090355
- [Result] Friesecke S, Trager K, Schittek GA, Molnar Z, Bach F, Kogelmann K, Bogdanski R, Weyland A, Nierhaus A, Nestler F, Olboeter D, Tomescu D, Jacob D, Haake H, Grigoryev E, Nitsch M, Baumann A, Quintel M, Schott M, Kielstein JT, Meier-Hellmann A, Born F, Schumacher U, Singer M, Kellum J, Brunkhorst FM. International registry on the use of the CytoSorb(R) adsorber in ICU patients : Study protocol and preliminary results. Med Klin Intensivmed Notfmed. 2019 Nov;114(8):699-707. doi: 10.1007/s00063-017-0342-5. Epub 2017 Sep 4. PMID 28871441
- [Result] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Result] Moreno R, Vincent JL, Matos R, Mendonca A, Cantraine F, Thijs L, Takala J, Sprung C, Antonelli M, Bruining H, Willatts S. The use of maximum SOFA score to quantify organ dysfunction/failure in intensive care. Results of a prospective, multicentre study. Working Group on Sepsis related Problems of the ESICM. Intensive Care Med. 1999 Jul;25(7):686-96. doi: 10.1007/s001340050931. PMID 10470572
- [Result] Hetz H, Berger R, Recknagel P, Steltzer H. Septic shock secondary to beta-hemolytic streptococcus-induced necrotizing fasciitis treated with a novel cytokine adsorption therapy. Int J Artif Organs. 2014 May;37(5):422-6. doi: 10.5301/ijao.5000315. Epub 2014 Apr 17. PMID 24811308
- [Result] Kogelmann K, Jarczak D, Scheller M, Druner M. Hemoadsorption by CytoSorb in septic patients: a case series. Crit Care. 2017 Mar 27;21(1):74. doi: 10.1186/s13054-017-1662-9. PMID 28343448
- [Result] David S, Thamm K, Schmidt BMW, Falk CS, Kielstein JT. Effect of extracorporeal cytokine removal on vascular barrier function in a septic shock patient. J Intensive Care. 2017 Jan 21;5:12. doi: 10.1186/s40560-017-0208-1. eCollection 2017. PMID 28127437
- [Result] Nemeth E, Kovacs E, Racz K, Soltesz A, Szigeti S, Kiss N, Csikos G, Koritsanszky KB, Berzsenyi V, Trembickij G, Fabry S, Prohaszka Z, Merkely B, Gal J. Impact of intraoperative cytokine adsorption on outcome of patients undergoing orthotopic heart transplantation-an observational study. Clin Transplant. 2018 Apr;32(4):e13211. doi: 10.1111/ctr.13211. Epub 2018 Feb 27. PMID 29377282
- [Result] Trasy D, Tanczos K, Nemeth M, Hankovszky P, Lovas A, Mikor A, Laszlo I, Hajdu E, Osztroluczki A, Fazakas J, Molnar Z; EProK study group. Early procalcitonin kinetics and appropriateness of empirical antimicrobial therapy in critically ill patients: A prospective observational study. J Crit Care. 2016 Aug;34:50-5. doi: 10.1016/j.jcrc.2016.04.007. Epub 2016 Apr 13. PMID 27288610
- [Result] Riedel S. Procalcitonin and the role of biomarkers in the diagnosis and management of sepsis. Diagn Microbiol Infect Dis. 2012 Jul;73(3):221-7. doi: 10.1016/j.diagmicrobio.2012.05.002. PMID 22704255
- [Result] Nylen ES, Whang KT, Snider RH Jr, Steinwald PM, White JC, Becker KL. Mortality is increased by procalcitonin and decreased by an antiserum reactive to procalcitonin in experimental sepsis. Crit Care Med. 1998 Jun;26(6):1001-6. doi: 10.1097/00003246-199806000-00015. PMID 9635646
- [Result] Schadler D, Pausch C, Heise D, Meier-Hellmann A, Brederlau J, Weiler N, Marx G, Putensen C, Spies C, Jorres A, Quintel M, Engel C, Kellum JA, Kuhlmann MK. The effect of a novel extracorporeal cytokine hemoadsorption device on IL-6 elimination in septic patients: A randomized controlled trial. PLoS One. 2017 Oct 30;12(10):e0187015. doi: 10.1371/journal.pone.0187015. eCollection 2017. PMID 29084247
- [Result] Trasy D, Molnar Z. Procalcitonin - Assisted Antibiotic Strategy in Sepsis. EJIFCC. 2017 May 1;28(2):104-113. eCollection 2017 May. PMID 28757818
- [Result] Pomare Montin D, Ankawi G, Lorenzin A, Neri M, Caprara C, Ronco C. Biocompatibility and Cytotoxic Evaluation of New Sorbent Cartridges for Blood Hemoperfusion. Blood Purif. 2018;46(3):187-195. doi: 10.1159/000489921. Epub 2018 Jun 8. PMID 29886501
- [Result] Ankawi G, Fan W, Pomare Montin D, Lorenzin A, Neri M, Caprara C, de Cal M, Ronco C. A New Series of Sorbent Devices for Multiple Clinical Purposes: Current Evidence and Future Directions. Blood Purif. 2019;47(1-3):94-100. doi: 10.1159/000493523. Epub 2018 Sep 25. PMID 30253409
- [Result] Rodriguez LE, Suarez EE, Loebe M, Bruckner BA. Ventricular assist devices (VAD) therapy: new technology, new hope? Methodist Debakey Cardiovasc J. 2013 Jan-Mar;9(1):32-7. doi: 10.14797/mdcj-9-1-32. PMID 23519193
- [Result] Lietz K, Long JW, Kfoury AG, Slaughter MS, Silver MA, Milano CA, Rogers JG, Naka Y, Mancini D, Miller LW. Outcomes of left ventricular assist device implantation as destination therapy in the post-REMATCH era: implications for patient selection. Circulation. 2007 Jul 31;116(5):497-505. doi: 10.1161/CIRCULATIONAHA.107.691972. Epub 2007 Jul 16. PMID 17638928
- [Result] Hetzer R, Delmo Walter EM. Trends and outcomes in heart transplantation: the Berlin experience. HSR Proc Intensive Care Cardiovasc Anesth. 2013;5(2):76-80. PMID 23888228
- [Result] Chen YF, Tsai WC, Lin CC, Tsai LY, Lee CS, Huang CH, Pan PC, Chen ML. Effect of leukocyte depletion on endothelial cell activation and transendothelial migration of leukocytes during cardiopulmonary bypass. Ann Thorac Surg. 2004 Aug;78(2):634-42; discussion 642-3. doi: 10.1016/j.athoracsur.2004.02.091. PMID 15276536

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT05042622/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-15): https://cdn.clinicaltrials.gov/large-docs/22/NCT05042622/ICF_001.pdf